CLINICAL TRIAL: NCT05135312
Title: Monitoring Nail Changes in Patients With Psoriatic Disease Treated With Etanercept Using Non- Invasive Optical Coherence Tomography
Brief Title: Etanercept Therapy for Nails Psoriasis Monitoring With Noninvasive Imaging
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: OptiSkin Medical (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Orit Markowitz MD, Chief Medical Ofiicer, OptiSkin Medical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTI-004
Record Dates: First submitted 2021-11-17; First posted 2021-11-26 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Psoriasis; Psoriatic Arthritis; Psoriatic Nail
Keywords: Psoriasis Nails; Psoriatic Arthritis; Enbrel; Biologic
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Etanercept; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Etanercept (Other): 50mg etanercept subcutaneously twice weekly for 3 months, followed by once weekly for another 3 months for a total duration of 6 months or 24 weeks.
  Interventions: Drug: Etanercept; Device: OCT

INTERVENTIONS:
Drug: Etanercept — TNF-alpha inhibitors improve nail psoriasis.
  Other Names: Enbrel
Device: OCT — Optical Coherence Tomography is a noninvasive imaging device that can be used to monitor nail disease severity.
  Other Names: Optical Coherence Tomography

SUMMARY:
OptiSkin is now enrolling a new study to monitor nail changes in patients with nail psoriasis treated with Enbrel® (etanercept) with optical coherence tomography (OCT).

DETAILED DESCRIPTION:
Psoriasis often affects the fingernails, making them yellow, brittle, painful and prone to infections. These symptoms can be difficult to manage, so OptiSkin is now enrolling a new study to monitor nail changes in patients with nail psoriasis treated with Enbrel® (etanercept) with optical coherence tomography (OCT).

OCT is being studied as a way to better diagnosis psoriatic nail disease, monitor response to therapy, and identify changes even before they become apparent, potentially leading to earlier treatment or prevention of future psoriatic arthritis.

Study-related care and medication are provided at no cost, and reimbursement for reasonable local transportation may be available to qualified individuals.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe psoriasis
* Psoriasis affecting the fingernails

Exclusion Criteria:

* Previous treatment with Enbrel® (etanercept)
* Active infection
* Rheumatoid arthritis
* Any personal or family history of any neurologic demyelinating disease
* Receipt of investigational drugs or "biologics" within 4 weeks of the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-08-08 (Estimated); Study Completion 2022-08-08 (Estimated)

PRIMARY OUTCOMES:
NAPSI | Baseline to 24 weeks
  Nail Psoriasis Severity Index (NAPSI) score is an established measure of nail disease ranging from 0-100. A higher score indicates more severe nails psoriasis.
OCT (clinical) | Baseline to 24 weeks
  Optical Coherence Tomography is noninvasive imaging that can be used to monitor nail disease severity.

SECONDARY OUTCOMES:
OCT (sub-clinical) | Baseline to 24 weeks
  Optical Coherence Tomography is noninvasive imaging that will be used to detect subclinical changes in otherwise healthy-appearing nails.
Dermoscopy | Baseline to 24 weeks
  Dermoscopy allows for the examination of the skin using skin surface microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Orit Markowitz, MD, Principal Investigator — OptiSkin Medical
Locations (1):
- OptiSkin Medical, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No